CLINICAL TRIAL: NCT03723850
Title: Effect of Noninvasive Electrical Brain Stimulation on Memory Performance at Different Times of Day in Younger and Older Adults
Brief Title: Effect of Noninvasive Electrical Brain Stimulation on Memory at Different Times of Day in Younger and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB18-1246; R21AG060444 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Effect of tDCS on Memory in Older and Younger Adults
Keywords: Transcranial Direct Current Stimulation; Memory; Prefrontal Cortex

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the participant, nor the research assistant administering tDCS will know if the participant is receiving active tDCS or sham tDCS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Older, active tDCS, dlPFC (Experimental): Older adults (ages 60-75) randomized to this arm will receive 2 sessions of active tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex. One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  2.
  Interventions: Device: Active tDCS
- Older, sham tDCS, dlPFC (Sham Comparator): Older adults (ages 60-75) randomized to this arm will receive 2 sessions of sham tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex. One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  Interventions: Device: Sham tDCS
- Younger, active tDCS, dlPFC (Experimental): Younger adults (ages 18-30) randomized to this arm will receive 2 sessions of active tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex. One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  Interventions: Device: Active tDCS
- Younger, sham tDCS, dlPFC/parietal (Sham Comparator): Younger adults (ages 18-30) randomized to this arm will receive 2 sessions of sham tDCS stimulation (Soterix Medical) delivered to either the left dorsolateral prefrontal cortex (area F3 using the 10-20 EEG system, n = 25), or the left parietal cortex (area P5 using the 10-20 EEG system, n = 25). One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  Interventions: Device: Sham tDCS
- Younger, active tDCS, parietal cortex (Active Comparator): Younger adults (ages 18-30) randomized to this arm will receive 2 sessions of active tDCS stimulation (Soterix Medical) delivered to the left parietal cortex (area P5 using the 10-20 EEG system). One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  Interventions: Device: Active tDCS

INTERVENTIONS:
Device: Active tDCS — The brain is stimulated for 20 minutes with mild electrical current (maximum 2 mA) with two 7 cm x 5 cm electrodes placed on the scalp, using a standard 1x1 tDCS Clinical Trials device (Soterix Medica, NY), specialized for double-blinding.
  Arms: Older, active tDCS, dlPFC; Younger, active tDCS, dlPFC; Younger, active tDCS, parietal cortex
Device: Sham tDCS — The brain is not stimulated for 20 minutes with mild electrical current, but instead a sham procedure is administered using a standard 1x1 tDCS Clinical Trials device (Soterix Medica, NY), specialized for double-blinding.
  Arms: Older, sham tDCS, dlPFC; Younger, sham tDCS, dlPFC/parietal

SUMMARY:
This study will investigate the extent to which tDCS to dorsolateral prefrontal cortex (or dlPFC) impacts memory performance as a function of time-of-day in younger and older adults.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) is the safest and most accessible, non-invasive brain stimulation technique available for testing causal links between different brain regions and functions, by manipulating cognitive abilities. By identifying key experimental factors that can improve the reliability and robustness of stimulation effects on cognitive performance in different age groups, this project should lead to the widespread adoption of these design features in future applications. This study will investigate the extent to which tDCS to dorsolateral prefrontal cortex (or dlPFC) impacts recollection accuracy and working memory performance as a function of time-of-day in younger and older adults. Moreover, this study will test the extent that tDCS to dlPFC impacts memory performance by impacting information-specific processes and/or cognitive control processes that operate across different types of information, thereby informing basic theories of how dlPFC contributes to memory in younger and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (according to the Edinburgh Handedness Inventory)
* Normal or corrected vision
* Fluent in English (started learning by age 6)
* Ability to understand and provide informed consent for study procedures, and to comply - with study procedures for the entire length of the study.
* For individuals in the 'younger adults' group, must be between 18 and 30 years of age
* For individuals in the 'older adults' group, must be between 60 and 75 years of age
* A score of 23 or above on the Montreal Cognitive Assessment (out of 30, education-corrected) is required. This is to minimize the inclusion of suspected mild cognitive impairment (MCI) or dementia, targeting individuals that score in the normal range according to the recent meta-analysis of MoCA's ability to differentiate normal aging from MCI in Carson et al. (2018, Int. J of Geriatric Psychiatry).
* Performance above threshold on the episodic memory task during the baseline session. The threshold is defined as having a hit rate that is at least 5% greater than the false alarm rate, where hit rate is defined as the number of studied items identified as studied, divided by the total number of studied items, and false alarm rate is defined as the number of new items identified as studied, divided by the total number of new items. We don't anticipate this threshold to exclude many, if any subjects.

Exclusion Criteria:

* Neuropsychological conditions associated with cognitive decline or seizure
* Cochlear implants or metal in the brain/skull (except titanium)
* Psychoactive medications, or diagnosis of depression, bipolar disorder, or any psychotic diagnoses
* History of excessive use (clinically treated) alcohol or narcotics
* Hospitalization for head trauma (e.g. concussions) in the past 5 years
* Individuals above a threshold score on an assessment of depression, specifically, a score of 10 or above on the Patient Health Questionnaire (PHQ-9)(Manea et al., 2012)
* Risk of pregnancy
* Low tolerance of skin irritation
* Prior brain stimulation experience (self-report)
* Ongoing cognitive or sensory deficits/symptoms from a previous (or current) COVID-19 infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Galllo, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will post data on the Open Science Framework (online), so that de-identified data will be made available to any outside researcher. Shared data will include, at a minimum, an excel data file used to summarize all participant cognitive data. Any computer scripts or stimuli used for task development also will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will become available within 6 months of publication of the relevant results.
Access Criteria: The investigators will use the Open Science Framework for making data available.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants have the right to end their participation at any time. In addition, the PI may terminate participation if a participant is in obvious non-compliance with the study procedures (e.g., responding randomly or sleeping during the cognitive task) or shows signs of moderate or severe adverse events associated with the study procedures (e.g., excessive discomfort with the tDCS electrodes). Enrolled participants may not continue in the study if they meet any of our exclusion criteria.
Groups:
- Older, Active tDCS, dlPFC: Older adults (ages 60-75) randomized to this arm will receive 2 sessions of active tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex. One session will occur in the morning (8 or 9am) and one will occur on a separate day in the afternoon (3 or 4pm).
  2.
  Active tDCS: The brain is stimulated for 20 minutes with mild electrical current (maximum 2 mA) with two 7 cm x 5 cm electrodes placed on the scalp, using a standard 1x1 tDCS Clinical Trials device (Soterix Medica, NY), specialized for double-blinding.
Period: Overall Study
Arm/Group | Older, Active tDCS, dlPFC | Older, Sham tDCS, dlPFC | Younger, Active tDCS, dlPFC | Younger, Sham tDCS, dlPFC/Parietal | Younger, Active tDCS, Parietal Cortex
Started | 49 | 45 | 54 | 52 | 51
Completed | 46 | 45 | 51 | 51 | 48
Not Completed | 3 | 0 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older, Active tDCS, dlPFC | Older, Sham tDCS, dlPFC | Younger, Active tDCS, dlPFC | Younger, Sham tDCS, dlPFC/Parietal | Younger, Active tDCS, Parietal Cortex | Total
Number analyzed (Participants) | 46 | 45 | 51 | 51 | 48 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 51 | 51 | 48 | 150
  >=65 years | 46 | 45 | 0 | 0 | 0 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.56 (4.58) | 67.06 (4.61) | 20.80 (2.90) | 20.90 (3.23) | 21.40 (3.06) | 39.54 (3.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 30 | 31 | 27 | 148
  Male | 15 | 16 | 21 | 20 | 21 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 9 | 11 | 14 | 38
  Not Hispanic or Latino | 40 | 38 | 41 | 38 | 34 | 191
  Unknown or Not Reported | 3 | 6 | 1 | 2 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 12 | 17 | 10 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 22 | 7 | 2 | 5 | 58
  White | 19 | 22 | 24 | 29 | 27 | 121
  More than one race | 5 | 1 | 6 | 1 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 51 | 51 | 48 | 241

OUTCOME MEASURES:

1. Primary Outcome: Episodic Memory Performance
Description: To measure episodic memory performance, participants will perform a recollection task. They will first study picture and word stimuli (encoding phase). On the subsequent memory test (retrieval phase), participants will be asked to differentiate between studied and non-studied items, as well as recollecting the previous format for studied items (i.e. recollecting the picture or word). For each tested item, participants will also be asked to make a confidence judgement about their response. The primary dependent variable (DV) will be the proportion of studied items attributed to the correct source minus the proportion of nonstudied items incorrectly attributed to that same source.
Time Frame: This task is performed immediately after tDCS is administered, and lasts approximately 20 minutes.
Population: Cognitively-normal adults.
Measure: Mean (Standard Deviation); unit: proportion of items
Arm/Group | Older, Active tDCS, dlPFC | Older, Sham tDCS, dlPFC | Younger, Active tDCS, dlPFC | Younger, Sham tDCS, dlPFC/Parietal | Younger, Active tDCS, Parietal Cortex
Number analyzed (Participants) | 46 | 45 | 51 | 51 | 48
proportion of items | 0.34 (0.25) | 0.32 (0.25) | 0.46 (0.26) | 0.50 (0.23) | 0.49 (0.24)

2. Secondary Outcome: Working Memory Performance
Description: To measure working memory performance, participants will perform two versions of the N-back task -- a verbal version (i.e., presenting the numbers 1-9 in a varied sequence) and a visuospatial version (i.e., presenting a colored square in one of 9 locations on a 3x3 grid in a varied sequence). The primary DV will be working memory accuracy: proportion of targets correctly identified minus the proportion of lures incorrectly endorsed.
Time Frame: This task lasts approximately 10 minutes and is performed immediately after the episodic memory task (approximately 20 minutes after the end of the tDCS session).
Population: cognitively-normal adults
Measure: Mean (Standard Deviation); unit: proportion of items
Arm/Group | Older, Active tDCS, dlPFC | Older, Sham tDCS, dlPFC | Younger, Active tDCS, dlPFC | Younger, Sham tDCS, dlPFC/Parietal | Younger, Active tDCS, Parietal Cortex
Number analyzed (Participants) | 44 | 43 | 47 | 48 | 42
proportion of items | 0.60 (0.31) | 0.60 (0.30) | 0.60 (0.26) | 0.58 (0.25) | 0.60 (0.26)

ADVERSE EVENTS:
Time Frame: The targeted timeframe was 7 to 12 days per participant, from baseline day to the final testing session.
Description: Does not differ. All adverse experiences will be recorded in the Adverse Events Survey . If the event is classified as a Serious Adverse Event, the PI will be notified immediately.
Arm/Group | Older, Active tDCS, dlPFC | Older, Sham tDCS, dlPFC | Younger, Active tDCS, dlPFC | Younger, Sham tDCS, dlPFC/Parietal | Younger, Active tDCS, Parietal Cortex
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/45 | 0/54 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/45 | 0/54 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 49/49 | 45/45 | 54/54 | 52/52 | 47/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older, Active tDCS, dlPFC (N=49) | Older, Sham tDCS, dlPFC (N=45) | Younger, Active tDCS, dlPFC (N=54) | Younger, Sham tDCS, dlPFC/Parietal (N=52) | Younger, Active tDCS, Parietal Cortex (N=51)
Non-Serious Adverse Events (Investigations) | 49 (49) | 45 (45) | 54 (54) | 52 (52) | 47 (47) — Any reported sensations participants felt (e.g., tingling/tickling, burning, discomfort, itching) around the stimulation site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03723850/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03723850/SAP_001.pdf